CLINICAL TRIAL: NCT00961064
Title: A Pilot Study of a Thrombopoietin-Receptor Agonist (TPO-R Agonist), Eltrombopag, in Patients With Low to Int-2 Risk Myelodysplastic Syndrome (MDS)
Brief Title: A Pilot Study of a Thrombopoietin-Receptor Agonist, Eltrombopag, in Patients With Low to Int-2 Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090199; 09-H-0199
Record Dates: First submitted 2009-08-15; First posted 2009-08-18 (Estimated); Results first posted 2019-08-22 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Myelodysplastic Syndromes; Thrombocytopenia
Keywords: Hematopoiesis; Thrombocytopenia; Autoimmunity; Megakaryocytes; Bone Marrow Fibrosis; Myelodysplastic Syndrome; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes; Thrombocytopenia; Autoimmune Diseases; Primary Myelofibrosis | interventions — eltrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eltrombopag in Low to Int-2 Risk Myelodysplastic Syndrome (MDS) (Experimental): Eltrombopag will be initiated at 50 mg/day (Asians 25 mg/day) and dose adjusted up to 150mg/day based response and safety in participants with Low to Int-2 Risk Myelodysplastic Syndrome (MDS)
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag will be initiated at 50 mg/day (Asians 25 mg/day) and dose adjusted up to 150mg/day based response and safety
  Other Names: PROMACTA

SUMMARY:
Background:

* Myelodysplastic syndromes (MDS) are bone marrow disorders characterized by anemia, neutropenia, and thrombocytopenia (low red blood cell, white blood cell, and platelet counts). Patients with MDS are at risk for symptomatic anemia, infection, and bleeding, as well as a risk of progression to acute leukemia. Standard treatments for MDS have significant relapse rates. MDS patients with thrombocytopenia who fail standard therapies require regular, expensive, and inconvenient platelet transfusions, and are at risk for further serious bleeding complications.
* Eltrombopag is a drug designed to mimic the protein thrombopoietin, which causes the body to make more platelets. Eltrombopag has been able to increase platelet counts in healthy volunteers and in patients with chronic ITP (a disease where patients destroy their own platelets very rapidly and thus develop thrombocytopenia), but researchers do not know if the drug can increase platelet counts in patients with MDS.

Objectives:

* To find out whether eltrombopag can improve platelet counts in patients with MDS.
* To determine whether eltrombopag is safe for patients with MDS.

Eligibility:

* Patients 18 years of age and older who have consistently low blood platelet counts related to MDS that has not responded to conventional treatment.
* Platelet count ≤ 30,000/μL or platelet-transfusion-dependence (requiring at least 4 platelet transfusions in the 8 weeks prior to study entry); OR hemoglobin less than 9.0 gr/dL or red cell transfusion-dependence (requiring at least 4 units of PRBCs in the eight weeks prior to study entry) OR ANC≤500

Design:

* Treatment with eltrombopag tablets once per day for 16-20 weeks.
* Participants will be monitored closely throughout the initial treatment, with weekly blood tests and separate evaluations at the National Institutes of Health (NIH) treatment center every 4 weeks. Bone marrow biopsies may be conducted to check for abnormalities in bone marrow.
* If patients show signs of improved platelet counts after 90 days, treatment will continue with additional doses of eltrombopag.
* Patients who discontinue taking eltrombopag will be evaluated at the NIH treatment center 4 weeks after ending treatment, and again 6 months after ending treatment to check for potential side effects.

DETAILED DESCRIPTION:
The myelodysplastic syndromes (MDS) are bone marrow disorders characterized by anemia, neutropenia, and thrombocytopenia. Patients with MDS are at risk for symptomatic anemia, infection, and bleeding, as well as a variable risk of progression to acute leukemia. With the exception of stem cell transplant, the standard treatments for MDS are rarely curative, and relapse rates are significant. MDS patients with cytopenias who fail standard therapies require regular blood or platelet transfusions which are expensive and inconvenient, and are at risk for serious bleeding complications.

Thrombopoietin (TPO) is the principal regulator of platelet production by megakaryocytes in the bone marrow. A 2nd generation TPO-agonist, eltrombopag (Promacta ) has been shown to increase platelets in thrombocytopenic patients with chronic immune thrombocytopenic purpura (ITP). Eltrombopag is administered orally, is well-tolerated, and is FDA approved for the treatment of thrombocytopenia in patients with chronic ITP who failed to respond to standard treatment.

Because the management of MDS patients with persistent cytopenias remains unsatisfactory and novel therapeutic approaches are needed, we propose a non-randomized, pilot, phase II study of eltrombopag in low to Int-2 risk MDS subjects with thrombocytopenia and anemia cytopenias who are either untreated or cytopenias that persist despite treatment with standard therapies to assess its utility in these settings.

Subjects will initiate study medication at an oral dose of 50 mg/day (25 mg/day for East Asians), which will be adjusted as clinically indicated to the lowest dose that maintains a stable platelet count greater than or equal to 20,000/microL above baseline while maximizing tolerability. Treatment response will be any increase in a cytopenia, in the lineage that fulfilled eligibility criteria for enrollment and will be defined as: (a) platelet count increases to 20,000/microL above baseline at 16 or 20 weeks , or stable platelet counts with transfusion independence for a minimum of 8 weeks in subjects who were previously transfusion dependent; (b) erythroid response for subjects with a pretreatment hemoglobin of less than 9 g/dL will be defined as an increase in hemoglobin by greater than or equal to 1.5g/dL without packed red blood cell (PRBC) transfusion support, or a reduction in the units of PRBC transfusions by at least 50% during the eight consecutive weeks prior to response assessment compared with the pretreatment transfusion number in the previous 8 weeks; (c) neutrophil response will be defined in those with a pretreatment absolute neutrophil count (ANC) of < 0.5 times 10(9)/L as at least a 100% increase or an absolute increase > 0.5 times 10(9)/L. Subjects meeting a response may remain on the extended access until they meet an off study criteria or the study is closed.

Subjects with response at 16 or 20 weeks may be consented for entry into the extended access part of the trial. In the event that a subject is transfused platelets for a count >10,000/microL without a medical indication during the study period, the subject may continue on study drug and the response assessment may be extended for an additional 4 weeks to week 20, at the discretion of the principal investigator. Subjects with evidence for a clinical response in any lineage at 16 weeks but not yet meeting full primary endpoint response criteria, and who are tolerating investigational treatment, may receive an additional 4 weeks of eltrombopag and be reassessed after 20 weeks. At that time, if they meet primary endpoint response criteria, they will be eligible to enter the extended access part of the study. If they do not meet primary endpoint response criteria, eltrombopag will be discontinued.

Primary objective is to assess the efficacy of eltrombopag in patients with low to Int-2 risk MDS. Safety of eltrombopag in this subject population will be assessed concurrently.

Secondary objectives include the toxicity profile of extended treatment with eltrombopag (treatment longer than 4 months), reduction in incidence and severity of bleeding episodes, and response following extended access to study drug (treatment longer than 4 months).

The primary endpoint will be the portion of drug responders as defined by changes in the platelet count and/or platelet transfusion requirements, or the proportion of subjects who meet erythroid response, or neutrophil response criteria.. Platelet response is defined as platelet count increases to 20,000/microL above baseline at 16 or 20 weeks, or stable platelet counts with transfusion independence for a minimum of 8 weeks. Erythroid response for subjects with a pretreatment hemoglobin of less than 9 g/dL will be defined as an increase in hemoglobin by greater than or equal to 1.5g/dL without packed red blood cell (PRBC) transfusion support, or a reduction in the units of PRBC transfusions by at least 50% during the eight consecutive weeks prior to response assessment compared with the pretreatment transfusion number in the previous 8 weeks. Neutrophil response will be defined in those with a pretreatment absolute neutrophil count (ANC) of <0.5 times 10(9)/L as at least a 100% increase or an absolute increase > 0.5 times 10(9)/L. Subjects with an erythroid, and/or neutrophil response at 16 weeks may continue study medication (extended access) until they meet an off study criteria. Subjects with erythroid, or neutrophil response at 16 weeks may continue study medication for an additional 4 weeks (to ensure eligibility) prior to being consented for entry into the extended access part of the trial. Patients may remain on the extended access until they met an off study criteria.

The toxicity profile will be measured using the CTCAE Version 4.0 criteria.

Secondary endpoints will include incidence of grade 2 or higher bleeding events as measured by CTCAE v. 4.0; changes in serum thrombopoietin level, measured at 4 months; and progression to higher risk MDS as measured by IWG criteria.

ELIGIBILITY:
* INCLUSION CRITERIA:

Diagnosis of MDS, with WHO classification of refractory anemia, refractory cytopenia with unilineage dysplasia (RCUD), RARS, RCMD-RS, or RCMD.

IPSS risk scores of low, intermediate-1, or intermediate-2.

Platelet count less than or equal to 30,000/ microL or platelet-transfusion-dependence (requiring at least 4 platelet transfusions in the 8 weeks prior to study entry); or hemoglobin less than 9.0 gr/dL or red cell transfusion-dependence (requiring at least 4 units of PRBCs in the eight weeks prior to study entry) OR ANC less than or equal to 500

Age greater than or equal to 18 years old

Treatment naive or off all other treatments for MDS (except stable dosing of filgrastim [G-CSF], erythropoietin, and transfusion support) for at least four weeks. G-CSF can be used before, during and after the protocol treatment for subjects with documented neutropenia (<500/UI) as long as they meet the criteria for other cytopenia as stated above. G-CSF must be held for 3 weeks prior to enrollment bone marrow biopsy and prior to each study assessment bone marrow biopsy, unless clinically indicated to avoid infections per PI discretion.

Adequate liver function, as evidenced by total serum bilirubin less than or equal to 1.5 times the upper limit of normal patients with Gilbert's disease are eligible, provided intermittent indirect hyperbilirubinemia, AST or ALT less than or equal to 5 times the upper limit of normal.

A serum creatinine concentration less than or equal to 2 times ULN

EXCLUSION CRITERIA:

WHO classification of chronic myelomonocytic leukemia (CMML), RAEB-1, RAEB-2, AML

Treatment with horse or rabbit ATG or Campath within 6 months of study entry

Subjects with liver cirrhosis including subjects infected with Hepatitis B or C

Subjects with HIV

Infection not adequately responding to appropriate therapy

History of malignancy treated with chemotherapy and cytogenetic abnormalities suggestive of secondary myelodysplasia.

Moribund status or concurrent hepatic, renal, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient s ability to tolerate protocol therapy

Life expectancy of less than 3 months

Hypersensitivity to eltrombopag or its components

Female subjects who are nursing or pregnant or are unwilling to take oral contraceptives or refrain from pregnancy if of childbearing potential

Unable to understand the investigational nature of the study or give informed consent or does not have a legally authorized representative or surrogate that can provide informed consent per section

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03-15 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal S Young, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kantarjian H, Giles F, List A, Lyons R, Sekeres MA, Pierce S, Deuson R, Leveque J. The incidence and impact of thrombocytopenia in myelodysplastic syndromes. Cancer. 2007 May 1;109(9):1705-14. doi: 10.1002/cncr.22602. PMID 17366593
- [Background] Houwerzijl EJ, Blom NR, van der Want JJ, Vellenga E, de Wolf JT. Megakaryocytic dysfunction in myelodysplastic syndromes and idiopathic thrombocytopenic purpura is in part due to different forms of cell death. Leukemia. 2006 Nov;20(11):1937-42. doi: 10.1038/sj.leu.2404385. Epub 2006 Sep 7. PMID 16990774
- [Background] Kalina U, Hofmann WK, Koschmieder S, Wagner S, Kauschat D, Hoelzer D, Ottmann OG. Alteration of c-mpl-mediated signal transduction in CD34(+) cells from patients with myelodysplastic syndromes. Exp Hematol. 2000 Oct;28(10):1158-63. doi: 10.1016/s0301-472x(00)00527-0. PMID 11027834
- [Derived] Giudice V, Feng X, Lin Z, Hu W, Zhang F, Qiao W, Ibanez MDPF, Rios O, Young NS. Deep sequencing and flow cytometric characterization of expanded effector memory CD8+CD57+ T cells frequently reveals T-cell receptor Vbeta oligoclonality and CDR3 homology in acquired aplastic anemia. Haematologica. 2018 May;103(5):759-769. doi: 10.3324/haematol.2017.176701. Epub 2018 Feb 1. PMID 29419434
- [Derived] Hosokawa K, Kajigaya S, Feng X, Desierto MJ, Fernandez Ibanez MD, Rios O, Weinstein B, Scheinberg P, Townsley DM, Young NS. A plasma microRNA signature as a biomarker for acquired aplastic anemia. Haematologica. 2017 Jan;102(1):69-78. doi: 10.3324/haematol.2016.151076. Epub 2016 Sep 22. PMID 27658437
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-H-0199.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Eltrombopag in Low to Int-2 Risk Myelodysplastic Syndrome (MDS): Eltrombopag (EPAG), a thrombopoietin receptor agonist, was started at 50 mg/day, up to a maximal dose of 150 mg/day, increasing the dose by 25mg every 2 weeks.
Period: Initial Treatment (Weeks 1 - 20)
Arm/Group | Eltrombopag in Low to Int-2 Risk Myelodysplastic Syndrome (MDS)
Started | 30
Completed | 14
Not Completed | 16
Not completed — No Response | 11
Not completed — Disease Progression | 3
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Period: Extended Access: Week 20 to Up to Year 5
Arm/Group | Eltrombopag in Low to Int-2 Risk Myelodysplastic Syndrome (MDS)
Started | 14
Completed | 7
Not Completed | 7
Not completed — Disease Progression | 3
Not completed — Lost Response | 1
Not completed — Non-compliant | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Eltrombopag in Low to Int-2 Risk Myelodysplastic Syndromes (MDS): Eltrombopag (EPAG), a thrombopoietin receptor agonist, was started at 50 mg/day, up to a maximal dose of 150 mg/day, increasing the dose by 25mg every 2 weeks.
Arm/Group | Eltrombopag in Low to Int-2 Risk Myelodysplastic Syndromes (MDS)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 19
  More than one race | 1
  Unknown or Not Reported | 2
Low Risk Myelodysplastic Syndromes (MDS) [Count of Participants; unit: Participants] — Low Risk Myelodysplastic Syndromes (MDS) are defined as having a low risk or a score of zero by the International Prognostic Scoring System (IPSS). A zero score is defined as: bone marrow blasts less than 5%, a good karyotype, and 1 of the following cytopenia: Hemoglobin < 10g/dL, Absolute neutrophil count < 1800/uL, Platelet count < 100,000/uL.
  IPSS score may range from zero which is the lowest score and is associated with better survival to a high score which is 3.5 and is associated with poorer survival when treatment is not provided.
  Participants | 2
Intermediate-1 Risk Myelodysplastic Syndromes (MDS) [Count of Participants; unit: Participants] — Intermediate-1 Risk Myelodysplastic Syndromes are defined as having low risk with score from 0.5 to 1 by the International Prognostic Scoring System (IPSS). A 0.5 to 1 score is defined as: bone marrow blasts 5 to 10%, intermediate to poor karyotype and 2 or 3 of the following: Hemoglobin < 10g/dL, Absolute neutrophil count < 1800/uL, Platelet count < 100,000/uL.
  IPSS score may range from zero which is the lowest score and is associated with better survival to a high score which is 3.5 and is associated with poorer survival when treatment is not provided.
  Participants | 27
Intermediate-2 Risk Myelodysplastic Syndromes (MDS) [Count of Participants; unit: Participants] — Intermediate-2 Risk Myelodysplastic Syndromes are defined as having a higher risk with score from 1.5 to 2 by the International Prognostic Scoring System (IPSS). A score of 1.5 to 2 is defined as: bone marrow blasts 11 to 30%, poor karyotype, and 2 or 3 of the following: Hemoglobin < 10g/dL, Absolute neutrophil count < 1800/uL, Platelet count < 100,000/uL.
  IPSS score may range from zero which is the lowest score and is associated with better survival to a high score which is 3.5 and is associated with poorer survival when treatment is not provided.
  Participants | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response Between Weeks 16 and 20
Description: The primary endpoint was hematologic response at 16 or 20 weeks, defined as either: (1) an increase in platelet counts =20.000/uL or transfusion independence for a minimum of 8 weeks; (2) hemoglobin (Hb) increase of =1.5g/dL from baseline, or a reduction in red blood cells (RBC) transfusion of at least 50%; or (3) an increase in absolute neutrophil counts (ANC) of =0.5x109/L or by at least 100% in patients with a baseline ANC <0.5x109/L.
Time Frame: 16 - 20 weeks
Population: The first 5 subjects enrolled were not counted toward the accrual target due to changes in protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Eltrombopag in Low to Int-1 Risk Myelodysplastic Syndrome (MDS): Eltrombopag (EPAG), a thrombopoietin receptor agonist, was started at 50 mg/day, up to a maximal dose of 150 mg/day, increasing the dose by 25mg every 2 weeks.
Arm/Group | Eltrombopag in Low to Int-1 Risk Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 25
Participants | 11

2. Secondary Outcome: Changes in Serum Thrombopoietin Level
Description: Changes in serum thrombopoietin level at 16 or 20 weeks
Time Frame: 16 - 20 weeks
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Eltrombopag in Low to Int-2 Risk Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 30
pg/mL | 2080 [71 to 4817]

3. Secondary Outcome: Number of Participants With Progression to Higher Risk Myelodysplastic Syndrome as Measured by International Working Group Criteria
Description: Number of participants with progression to higher risk Myelodysplastic syndrome (MDS) as measured by International Working Group (IWG) 2006 criteria in participants With Low to Int-2 Risk Myelodysplastic Syndrome (MDS) following Eltrombopag.
  Progression of disease per modified IWG criteria 2006 were considered: if patients with baseline bone marrow blasts of < 5% increase by ≥ 50% to >5% blasts; and either at least 50% decrease in granulocytes or platelets from maximum response, decreasing in Hb by 2g/dL or transfusion dependence. The acquisition of new cytogenetic abnormality without meeting other IWG criteria for progression was not considered disease progression.
Time Frame: up to 5 years
Population: intention to treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag in Low to Int-2 Risk Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 30
Participants | 6

4. Secondary Outcome: Number of Participants Who Achieved a Robust Response and Discontinued Eltrombopag
Description: Number of participants who achieved a robust response and discontinued Eltrombopag in extended access
  A robust response is defined as: as platelets >50,000/μL, hemoglobin > 10 g/dL in the absence of transfusions, and neutrophils > 1,000 for more than 8 weeks.
Time Frame: up to 5 years
Population: Analysis included those participants that participated in extended access portion of study
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag in Low to Int-1 Risk Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 14
Participants | 10

5. Secondary Outcome: Number of Participants With Grade 2 or Higher Bleeding Events Defined by Common Terminology Criteria for Adverse Events v. 4.0
Description: Number of Participants with Grade 2 or Higher Bleeding Events defined by Common Terminology Criteria for Adverse Events (CTCAE) v. 4.0.
  The NCI CTCAE is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline. Grade 1 Mild is asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 is moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL)*. Grade 3 is severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL**. Grade 4 if life-threatening consequences; urgent intervention indicated. Grade 5 is death related to AE.
Time Frame: up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag in Low to Int-2 Risk Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 30
Participants | 5

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Any observed or volunteered adverse events that are as listed in the Eltrombopag Package Insert and/or Investigator's Brochure will not be reported unless (1) the adverse event was not present at baseline exam; (2) the adverse event is previously unknown (not on the label); (3) the adverse event is more severe than on the label; (4) the frequency of the adverse events increases above the listed frequency; or (5) meets the criteria for a serious adverse event.
Arm/Group | Eltrombopag in Low to Int-2 Risk Myelodysplastic Syndrome (MDS)
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 12/30
Other Adverse Events (participants affected / at risk) | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag in Low to Int-2 Risk Myelodysplastic Syndrome (MDS) (N=30)
Death (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Investigation (Investigations) | 1
Nervous system disorder (Nervous system disorders) | 1
Bladder mass (Renal and urinary disorders) | 1
Hospitalisation (Surgical and medical procedures) | 10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag in Low to Int-2 Risk Myelodysplastic Syndrome (MDS) (N=30)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Jaundice (Blood and lymphatic system disorders) | 4
Ocular icterus (Blood and lymphatic system disorders) | 4
Petechiae (Blood and lymphatic system disorders) | 3
Dizziness (Cardiac disorders) | 7
Dyspnoea (Cardiac disorders) | 6
Oedema peripheral (Cardiac disorders) | 2
Blepharospasm (Eye disorders) | 2
Vision blurred (Eye disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 6
Faeces discoloured (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Gingival bleeding (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 6
Oropharyngeal pain (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 3
Chills (General disorders) | 2
Fatigue (General disorders) | 11
Flank pain (General disorders) | 2
Oedema (General disorders) | 3
Pain (General disorders) | 3
Pyrexia (General disorders) | 2
Bronchitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 4
Haemoglobin decreased (Investigations) | 9
Liver function test increased (Investigations) | 3
Neutrophil count decreased (Investigations) | 7
Platelet count decreased (Investigations) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Aphasia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 6
Insomnia (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Chromaturia (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 4
Skin discolouration (Skin and subcutaneous tissue disorders) | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 5
Sinus operation (Surgical and medical procedures) | 2

LIMITATIONS AND CAVEATS:
The first five participants enrolled were entered when eligibility criteria included only thrombocytopenia. They were not included in the efficacy analysis set, as requested by the Institutional Review Board, but were included for secondary endpoint and sensitivity analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT00961064/Prot_SAP_000.pdf